CLINICAL TRIAL: NCT02569528
Title: ImplemeNtation oF demOnstration pRoject for Health systeMs: Atrial Fibrillation (INFORM-AF) Part 1
Acronym: INFORM-AF
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Boehringer Ingelheim (Industry); Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00059115
Record Dates: First submitted 2015-10-05; First posted 2015-10-06 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; anticoagulation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients: Patients of consenting providers will complete a short survey and interview.
- Providers: Physicians treating patients with atrial fibrillation will complete a short survey and interview.

SUMMARY:
The goal of this study is to learn about the patient and provider perceptions, priorities, preferences, and willingness to use/prescribe anticoagulation as a stroke prevention therapy in patients with atrial fibrillation. Qualitative interviews will be performed with atrial fibrillation patients and providers caring for atrial fibrillation patients. The investigators want to understand the factors that influence decision-making about anticoagulation medications, and to gain insight into patients' and providers' knowledge of the risk of stroke and bleeding associated with oral anticoagulation. This feedback will help provide better education to providers caring for patients with atrial fibrillation and better care to patients with atrial fibrillation by developing tools to optimize the appropriate use of oral anticoagulation for patients with atrial fibrillation.

ELIGIBILITY:
Patient Inclusion Criteria:

1. adult patient age 18 or older;
2. English speaking;
3. diagnosed atrial fibrillation;
4. at least 1 risk factor for congestive heart failure, hypertension, age, diabetes, stroke (CHADS2) or 2 risk factors for CHADS2 with vascular disease, age, and sex (CHADS2-VASc) ;
5. no documented cognitive impairment per the medical record;
6. not being prescribed an oral anticoagulant

Provider Inclusion Criteria:

1. physician at one of the study sites treating patients diagnosed with atrial fibrillation

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will include 100 patients and 10 physicians, who are caring for those patients in the outpatient setting.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2015-10; Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Perceptions of using anticoagulation as a stroke prevention therapy in atrial fibrillation, as measured by survey and interview | one hour
  Each telephone interview (data collection time point) will be approximately one hour

SECONDARY OUTCOMES:
Willingness to use anticoagulation as a stroke prevention therapy in atrial fibrillation, as measured by survey and interview | one hour
  Each telephone interview (data collection time point) will be approximately one hour
preferences for using anticoagulation as a stroke prevention therapy in atrial fibrillation, as measured by survey and interview | one hour
  Each telephone interview (data collection time point) will be approximately one hour
priorities for using anticoagulation as a stroke prevention therapy in atrial fibrillation, as measured by survey and interview | one hour
  Each telephone interview (data collection time point) will be approximately one hour

CONTACTS AND LOCATIONS:
Overall Officials: Bradi B Granger, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Health System, Durham, North Carolina, United States